CLINICAL TRIAL: NCT02921672
Title: Feasibility Trial of a Mediterranean Diet Pattern to Prevent Cognitive Decline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003894; P30AG035982 (NIH)
Record Dates: First submitted 2016-09-29; First posted 2016-10-03 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Alzheimer's Disease; Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitively Normal (Active Comparator): Persons who are considered to have normal cognitive function. A registered dietician will meet with each person to discuss the Mediterranean Diet.
  Interventions: Other: Mediterranean Diet
- Mild Cognitive Impairment (Active Comparator): Persons diagnosed mild cognitive impairment (MCI). A registered dietician will meet with each person to discuss the Mediterranean Diet.
  Interventions: Other: Mediterranean Diet
- Mild to Moderate Alzheimer's Disease (Experimental): Persons diagnosed with mild to moderate Alzheimer's disease (AD). A registered dietician will meet with each person to discuss the Mediterranean Diet.
  Interventions: Other: Mediterranean Diet

INTERVENTIONS:
Other: Mediterranean Diet — Diet consisting of fruits, vegetables, grains, dairy, olive oils, seafood, and nuts. It is low in red meat and solid fats.

SUMMARY:
By doing this study, researchers hope to learn if older adults with and without cognitive impairment can adhere to a Mediterranean diet.

DETAILED DESCRIPTION:
Participants will be given instruction on following the study designed Mediterranean diet. Participation in the study will last about 9 weeks. Each person will be asked to follow the study diet for 6 weeks. During the study, participants will be asked to track the food they eat and will be monitored by a registered dietitian.

Potential participants need to be located within the KC metro area.

ELIGIBILITY:
Inclusion Criteria:

* Cognitively normal older adults over the age of 65 or individuals with a diagnosis of MCI or AD (any age)
* Have a study partner, if diagnosed with MCI or AD
* Body mass index (BMI) range between 20 - 35 kg/m2
* Speak English as a primary language

Exclusion Criteria:

* Serious medical risk
* Adherence to specialized diet regimes
* Already consume a Mediterranean diet pattern

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03; Primary Completion 2018-06-22 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Number of participants completing the study | Week 6
  Determine feasibility of this patient population's ability to maintain the diet. Outcome will be measured by the number of participants who complete the entire study.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah K Sullivan, PhD, RD, LD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No